CLINICAL TRIAL: NCT06288802
Title: Study of Wilms Tumors Among Patients of Shefa Al-Orman Children Cancer Hospital
Status: Recruiting | Type: Observational
Sponsor: South Egypt Cancer Institute (Other)
Collaborators: Shefa Al-orman Children Cancer Hospital (Unknown); Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Motaz Elzembely, Lecturer of Pediatric Hematology Oncology, South Egypt Cancer Institute
Other Study IDs: 04-2023-200647
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Wilms Tumor
Keywords: wilms; incidence; outcome
MeSH Terms: conditions — Wilms Tumor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross sectional observational study is to determine the percentage of Wilms tumors among pediatric cancers at Shefa Al-Orman Children Cancer Hospital from june 2020 to june 2024,to study the outcome of patients with Wilms tumor treated according to SIOP Umbrella protocol during the study period and to study the treatment related complications during therapy according to common terminology criteria of adverse events version 5.0 (CTCAE Version 5.0).

DETAILED DESCRIPTION:
Research Design and Methods:

Study design: cross sectional study Study setting: Shefa Al-Orman Children Cancer hospital Study period: from June 2020 to June 2024

Study Objectives:

1. To determine the percentage of Wilms tumors among pediatric cancers.
2. To study the outcome of patients with Wilms tumor treated according to SIOP Umbrella protocol (1).
3. To study the treatment related complications during therapy according to common terminology criteria of adverse events version 5.0 (CTCAE Version 5.0) (2).

Data collection: Each patient is subjected to all the following according to the centre policy:

I. History and physical examination at presentation:

1. Demographic data as: Age, sex, residence and date of diagnosis.
2. Clinical history and Physical examination including

   * Initial signs and symptoms of pediatric renal tumors including palpable abdominal mass, abdominal pain, hypertension, hematuria, weight loss, constipation, diarrhea, urinary tract infection, previous trauma….etc.
   * Associated congenital anomalies including. Aniridia, genitourinary anomalies, hemihypertrophy
   * Family history of cancer

II. Laboratory studies done for diagnosis of renal tumors at presentation:

- Complete blood count: presence/absence of polycythemia, anemia, thrombocytopenia

* Serum chemistries: blood urea nitrogen, creatinine, uric acid, Alanin transaminases, aspartate aminotransferase, serum bilirubin.
* Assessment of coagulation factors: prothrombin time, partial thromboplastin time

III. Imaging Studies:

1. Abdominal ultrasound
2. Abdominal CT scan or MRI with special attention to

   * Presence and function of the opposite kidney

   *Evidence of bilateral lesions

   *Evidence of involvement of renal vein or inferior vena cava with tumor

   *Lymph node involvement

   *Liver metastasis
3. Chest computed tomography scan.
4. Echocardiography: To

   * Assess myocardial contractility before starting cardiotoxic chemotherapy.
   * Detect the presence of tumor in the inferior vena cava or right atrium

IV. Pathology:

1. Ultrasound or CT guided True cut needle biopsy is indicated in the following conditions:

   A- Unusual clinical presentations:

   - Age > 5-6 years or less than 6 months

   B- Unusual findings by imaging:

   - Calcification

   - Voluminous adenopathies

   - Renal parenchyma not visible

   - Almost totally extrarenal process

   C- Contraindications for the use of Needle Biopsy:
   * Suspicion of rupture or hemorrhage
   * Needle biopsy is unlikely to be of benefit in pure cystic structures with no solid component. Immediate surgery to establish the diagnosis is recommended in such cases.

   V. Reporting of treament related complications include:

   Chemotherapy toxicity will be determined according to WHO Common Terminology Criteria for Adverse Events (CTCAE Version 5.0, 2017) (2).

   VI. Treatment: Patients are treated according to SIOP Umbrella protocol (1)

ELIGIBILITY:
Inclusion Criteria:

* Children and young adolescene younger than 18 years of age admitted and treated at Shefa Al-orman Children Cancer Hospital during the study period

Exclusion Criteria:

* Patients aged older than 18 years old, died early at presentation before starting chemotherapy, patients with non-Wilms renal tumors, relapsed renal tumors.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adolescene younger than 18 years of age admitted and treated at Shefa Al-orman Children Cancer Hospital during the study period
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall-survival (OS) | from date of diagnosis to last date of follow up or date of death for any cause
  will be calculated from date of diagnosis to last date of follow up or date of death for any cause

SECONDARY OUTCOMES:
Event-free survival (EFS) | the date of Wilms tumor diagnosis to the first treatment failure or date of last follow-up. Treatment failure included abandonment of treatment, death, and progressive or relapsed disease.
  will be measured from the date of Wilms tumor diagnosis to the first treatment failure or date of last follow-up. Treatment failure included abandonment of treatment, death, and progressive or relapsed disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elzembely, MD, Principal Investigator — South Egypt Cancer Institute
Locations (1):
- Shefa Al-orman Children Cancer Hospital, Luxor, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E, Becker C, Rogak LJ, Schrag D, Reeve BB, Spears P, Smith ML, Gounder MM, Mahoney MR, Schwartz GK, Bennett AV, Mendoza TR, Cleeland CS, Sloan JA, Bruner DW, Schwab G, Atkinson TM, Thanarajasingam G, Bertagnolli MM, Dueck AC. Composite grading algorithm for the National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Clin Trials. 2021 Feb;18(1):104-114. doi: 10.1177/1740774520975120. Epub 2020 Dec 1. PMID 33258687
- [Result] van den Heuvel-Eibrink MM, Hol JA, Pritchard-Jones K, van Tinteren H, Furtwangler R, Verschuur AC, Vujanic GM, Leuschner I, Brok J, Rube C, Smets AM, Janssens GO, Godzinski J, Ramirez-Villar GL, de Camargo B, Segers H, Collini P, Gessler M, Bergeron C, Spreafico F, Graf N; International Society of Paediatric Oncology - Renal Tumour Study Group (SIOP-RTSG). Position paper: Rationale for the treatment of Wilms tumour in the UMBRELLA SIOP-RTSG 2016 protocol. Nat Rev Urol. 2017 Dec;14(12):743-752. doi: 10.1038/nrurol.2017.163. Epub 2017 Oct 31. PMID 29089605